CLINICAL TRIAL: NCT06242990
Title: Developing and Feasibility Testing the Youth - Physical Activity Towards Health Intervention in Post-primary Schools in Northern Ireland
Brief Title: The Youth - Physical Activity Towards Health Intervention in Northern Ireland
Acronym: Y-PATH NI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Ulster (Other)
Collaborators: Northern Ireland Chest Heart and Stroke (Other); Dublin City University (Other); University College Cork (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: REC/23/0045
Record Dates: First submitted 2023-11-29; First posted 2024-02-05 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-01

CONDITIONS: Physical Inactivity
Keywords: Physical Activity; Physical Education; Children; Adolescents
MeSH Terms: conditions — Sedentary Behavior; Motor Activity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Y-PATH Intervention Group (Experimental): Participants will receive the Y-PATH NI intervention programme which is an adapted form of physical education classes.
  Interventions: Behavioral: Y-PATH NI
- Control Group (No Intervention): Participants will continue to receive their usual physical education classes.

INTERVENTIONS:
Behavioral: Y-PATH NI — The Y-PATH NI intervention provides a whole of school approach with student, teacher, parent and guardian components. Student components: Y-PATH resources delivered by physical education teachers (6 lesson plans, resource cards to use as teaching prompts), student handbook. Posters are also displayed in the sports hall/ PE department.
  Teacher components: Teachers will receive online and in-person training to deliver the Y-PATH programme. This component also targets all non-specialist PE teachers and includes workshops, information leaflets, development of a physical activity promotion charter and a step challenge.
  Parent/guardian components: Information session and leaflets distributed across the intervention period.
  Arms: Y-PATH Intervention Group

SUMMARY:
The Y-PATH programme is an evidence-based intervention programme that has been found to be successful at increasing levels of physical activity in school children in the Republic of Ireland. The Irish Heart Foundation collaborated with Dublin City University and University College Cork to disseminate the programme nationally. The intervention programme aims to improve physical activity levels of adolescents through education about the importance of physical activity for health and the development of fundamental movement skills, which are basic movements associated with physical activity, such as, catching, throwing, and running. The main aims of the Y-PATH NI study are:

* To explore Y-PATH as an intervention 'template', to lead the development of a research-informed model suitable for feasibility testing in a Northern Ireland context (Y-PATH NI).
* To undertake feasibility testing of the Y-PATH NI multi-component intervention aimed at increasing moderate-to-vigorous physical activity in 11-14 year olds.
* To conduct a process evaluation to determine primarily fidelity, but also acceptance and sustainability of the Y-PATH NI intervention.

ELIGIBILITY:
Inclusion Criteria:

Schools

* Post-primary schools in NI with at least one Year 8 class group commencing in the academic year 2023 will be eligible to take part in the study.
* Schools must have a minimum of one PE period/week timetabled for incoming Year 8 pupils,
* have an indoor sports hall (to facilitate intervention delivery)
* employ a qualified PE teacher (with at least 1 years' experience) to teach PE to the Year 8 class group.

Pupils

• All pupils (male and female) in the Year 8 classes identified by the school, who can take part in PE classes, will be eligible to participate in the study.

Teachers

* Male and female school staff
* PE specialist teachers (with at least 1 years' experience)
* Staff need to be over 18 years old.

Parents/Guardians

* Male and female parents/guardians
* aged over 18 years old
* with at least one child participating in the Y-PATH NI intervention.

Exclusion Criteria:

Schools

* Primary schools
* Schools which do not provided a minimum of one PE period/week timetabled for incoming Year 8 pupils,
* Schools without an indoor sports hall (to facilitate intervention delivery)
* Schools that do not employ a qualified PE teacher (with at least 1 years' experience) to teach PE to the Year 8 class group.

Pupils

* Pupils in Year 9 and above
* Pupils who do not take part in PE class (determined by the school)

Teachers

• Teachers not involved with the Y-PATH NI intervention

Parents/Guardians

• Not having at least one child who participated in the Y-PATH NI intervention

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 400 (Estimated)
Dates: Start 2024-02-23 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
The feasibility of recruiting schools/teachers to take part in the study | During recruitment phase, 1-2 months
  Ability to recruit schools/teachers to take part in the study. The research team will record the number of schools invited to take part and the number of schools who agree to participate in the study.
The feasibility of recruiting pupils to take part in the study | During recruitment phase, 1-2 months
  The research team will record the number of pupils who are invited to take part in each of the schools and the number of pupils who are recruited.
The feasibility of training the teachers | After baseline assessments have been completed, up to 2 months
  The number of teachers trained will be recorded and teachers complete an evaluation questionnaire to share their opinions on the training.
The feasibility of delivering Y-PATH NI in schools | Mid-point and end of study, up to 11 months in total
  Ability to deliver the intervention per protocol within schools. An intervention fidelity checklist will be completed as part of the process evaluation that will be carried out. The following questions will be included, Were all six Health related activity lesson plans delivered? Did teachers use the digital resources? Did teachers use the resource cards?
Acceptability of the Y-PATH NI Intervention to the pupils - self-report measure | Completed at the mid-point of the study (approximately 3-4 months after baseline)
  Pupils who are allocated to the intervention group will complete a self-report evaluation questionnaire which will ask for their opinions on the study (i.e. whether they enjoyed the study and if they were satisfied with the various components of the study). The scales will range from strongly disagree (1) to strongly agree (5).
Acceptability of the Y-PATH NI Intervention to the pupils - focus groups | Completed at the mid-point of the study (approximately 3-4 months after baseline)
  A sub-sample of pupils will participate in focus groups. The focus group would include 5-8 pupils and will aim to gather views and opinions on the Y-PATH NI intervention. A topic guide has been created for this focus group
Acceptability of the Y-PATH NI Intervention to the teachers | Completed at the mid-point of the study (approximately 3-4 months after baseline) and at the end of the study ( up to 11 months after baseline)
  Teachers will be asked to participate in an interview at the mid-point of the study and at the end of the study to share their opinions on the Y-PATH NI intervention. A topic guide will be used to guide the interview.
Acceptability of the Y-PATH NI Intervention to the teachers | Completed at the mid-point of the study (approximately 3-4 months after baseline)
  Teachers will be asked to complete a questionnaire at the mid-point of the study which asks questions about the acceptability of the intervention. Higher scores will indicate greater acceptability.
Acceptability of the Y-PATH NI Intervention to parents/guardians | Completed at the end of the study, up to 11 months after baseline.
  Parents of pupils who participated in the Y-PATH NI intervention will be invited to take part in an interview at the end of the study to gather their views on the Y-PATH NI intervention.

SECONDARY OUTCOMES:
Time spent in total physical activity, light physical activity, moderate-to-vigorous physical activity and sedentary behaviour | Measured at baseline, mid point (approximately 3- 4 months after baseline) and at the final follow up (up to 11 months after baseline measurement)
  Time spent in total physical activity, light physical activity, moderate-to-vigorous physical activity and sedentary behaviour, as measured by accelerometry
Body Mass Index | Measured at baseline, mid point (approximately 3- 4 months after baseline) and at the final follow up (up to 11 months after baseline measurement
  Weight (in kilograms) and height (in metres) will be measured at three time points throughout the study and body mass index will be calculated. Weight and height will be combined to report BMI in kg/m^2).
Proportion of participants meeting physical activity guidelines | Measured at baseline, mid point (approximately 3- 4 months after baseline) and at the final follow up (up to 11 months after baseline measurement
  Proportion of participants meeting physical activity guidelines determined by self-report questionnaire and accelerometry.
Enjoyment of physical education | Measured at baseline, mid point (approximately 3- 4 months after baseline) and at the final follow up (up to 11 months after baseline measurement
  Enjoyment of physical education will be measured using the Factors Influencing Enjoyment of Physical Education Enjoyment (FIPE) scale (Motl et al. 2001). This scale consists of 12 items on a 5-point Likert scale ranging from 1 (dislike a lot) to 5 (enjoy a lot) (range 12 - 60).
Experiences of physical education | Measured at baseline, mid point (approximately 3- 4 months after baseline) and at the final follow up (up to 11 months after baseline measurement
  Experiences of physical education will be assessed using a twelve item scale (e.g., I feel the activity I do in my PE class I do very well), with pupils indicating the extent to which they agree with the statement, from 'I don't agree at all' to I completely agree' (Woods et al. 2010). In line with previous research, a cut-off point of 36 will be used to distinguish between negative and positive experiences of PE (Clarke, 2019).
Self-efficacy for exercise | Measured at baseline, mid point (approximately 3- 4 months after baseline) and at the final follow up (up to 11 months after baseline measurement
  Self-efficacy will be assessed using the eight-item scale (e.g., I could exercise even if I was tired), with pupils indicating the extent to which the statement is 'very true' to 'not at all true' on a scale of 1 to 4. An average of the eight items gives an overall self-efficacy score between 1 (low self-efficacy) and 4 (high self-efficacy) (Garcia et al. 1998). This instrument has been used in this population previously, including the FifeActive survey (Rowe and Murtagh, 2012).
Physical self-confidence | Measured at baseline, mid point (approximately 3- 4 months after baseline) and at the final follow up (up to 11 months after baseline measurement
  The Physical Self-Confidence Scale will be used to assess the self-reported confidence in the adolescents ability to do 15 fundamental movement skills. Each of the skills will be rated on a scale from 1 -10, with 1 indicating no confidence and 10 indicating the participant is 'very confident' at performing each skill.
Behavioural Regulations in Exercise | Measured at baseline, mid point (approximately 3- 4 months after baseline) and at the final follow up (up to 11 months after baseline measurement
  The Behavioural Regulations in Exercise questionnaire (BREQ-3) will be used to assess reasons why participants take part in exercise and motivation to take part in exercise. Participants will be asked to rate each item on a scale from 0 (not true for me) to 4 (very true for me). A mean score will be calculated for each of the subscales included in this questionnaire: amotivation, external regulation, introjected regulation, identified regulation, integrated regulation and intrinsic regulation.
Screen time | Measured at baseline, mid point (approximately 3- 4 months after baseline) and at the final follow up (up to 11 months after baseline measurement.
  Screen time will be assessed using a one item tool, with participants asked to report the total number of hours and minutes per day engaged in screen time over the past week (Moore et al, 2020).

CONTACTS AND LOCATIONS:
Overall Officials: Angela Carlin, PhD, Principal Investigator — Ulster University
Locations (1):
- Ulster University, Londonderry, United Kingdom

IPD SHARING:
Plan to Share IPD: No